CLINICAL TRIAL: NCT03843151
Title: Relative Bioavailability of a Single Oral Dose of BI 1358894 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects (an Open-label, Fixed Sequence Study)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of BI 1358894 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0007; 2018-004274-10 (EudraCT Number)
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total of the 2-treatment, 2-period, fixed-sequence trial (Experimental): Treatment period 1 (Reference (R)): Oral administration of single dose of 10 milligram (mg) BI 1358894 (2 tablets of 5 mg) with 240 milliliter (mL) of water after an high-fat, high-calorie breakfast on Day 1 of Treatment Period 1.
  Treatment period 2 (Test (T)): Oral administration of 200 mg itraconazole (20 mL of 10 mg/mL solution) with 240 mL of water after an overnight fast for at least 10 h once daily for 14 days on Days -3 to 11 combined with a single dose of 10 mg BI 1358894 (2 tablets of 5 mg) on Day 1 of Treatment Period 2, 1.5 hours after administration of itraconazole.
  Administrations of BI 1358894 were separated by a washout interval of at least 17 days.
  Interventions: Drug: BI 1358894; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 1358894 — Oral administration of single dose of 10 milligram (mg) BI 1358894 (2 tablets of 5 mg) with 240 milliliter (mL) of water after an high-fat, high-calorie breakfast on Day 1 of Treatment Period 1.
Drug: Itraconazole — Oral administration of 200 mg itraconazole (20 mL of 10 mg/mL solution) with 240 mL of water after an overnight fast for at least 10 h once daily for 14 days on Days -3 to 11 combined with a single dose of 10 mg BI 1358894 (2 tablets of 5 mg) on Day 1 of Treatment Period 2, 1.5 hours after administration of itraconazole.

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 1358894 in plasma when given as oral single dose together with multiple oral doses of itraconazole (Test, T) as compared to when given alone as oral single dose (Reference, R).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active must use adequate contraception with their female partner throughout the study and until 1 month after the last administration of trial medication. Adequate methods are:

  * Sexual abstinence or
  * A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success) or
  * Surgical sterilisation (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner or
  * The use of condoms, if the female partner uses an adequate contraception method in addition, e.g., intrauterine device (IUD), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g. diaphragm with spermicide) Unprotected sexual intercourse with a female partner is not allowed throughout the study and until 1 month after the last administration of trial medication.

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* C-reactive protein (CRP)> Upper limit of normal (ULN), Erythrocyte sedimentation rate (ESR)≥15 millimeters/h, liver or kidney parameter above ULN, or any other laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medications or their excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Any lifetime history of suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
* Any suicidal ideation of type 2 to 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) in the past 12 months (i.e. active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
* Any history of drug-induced liver failure.
* History of ventricular dysfunction or congestive heart failure.
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed as an open-label, 2-treatment, 2-period, fixed sequence trial in healthy male subjects. Each subject was allocated to the same treatment sequence (Reference (R)-Test (T)).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Total of the 2-treatment, 2-period, Fixed-sequence Trial
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were treated with at least 1 dose of trial drug.
Arm/Group | Total of the 2-treatment, 2-period, Fixed-sequence Trial
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 Extrapolated to Infinity
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Data presented come from an analysis of variance (ANOVA) model on the logarithmic scale, this model included effects accounting for 'subject' and 'treatment'. The 'subject' effect was considered as random, whereas the 'treatment' effect was considered as fixed.
Time Frame: For each period: within 2.5 hours prior and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 7, 8, 10, 12, 16, 24, 34, 48, 72, 96, 120, 144, 168, 192, 216, 240, 312 and 480* hours after administration of BI 1358894. *only in the second period.
Population: Pharmacokinetic parameter analysis set (PKS) included all subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetic (PK) or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles*Hour per Liter
Groups:
- BI 1358894 + Itraconazole: Oral administration of 200 mg itraconazole (20 mL of 10 mg/mL solution) with 240 mL of water after an overnight fast for at least 10 h once daily for 14 days on Days -3 to 11 combined with a single dose of 10 mg BI 1358894 (2 tablets of 5 mg) on Day 1 of Treatment Period 2, 1.5 hours after administration of itraconazole.
Arm/Group | BI 1358894 | BI 1358894 + Itraconazole
Number analyzed (Participants) | 16 | 16
Nanomoles*Hour per Liter | 1623.89 (NA) — Geometric standard error = 1.07 | 3128.75 (NA) — Geometric standard error = 1.08
Statistical Analysis 1: Comparison: BI 1358894 vs BI 1358894 + Itraconazole; The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for 'subject' and 'treatment'. The 'subject' effect was considered as random, whereas the 'treatment' effect was considered as fixed; Test type: Other; Ratio = 192.67, 90% CI 2-sided [175.19 to 211.89] — The effect of itraconazole on BI 1358894 is estimated by the ratio of geometric mean (BI 1358894 + itraconazole / BI 1358894). geometric coefficient of variation (gCV) [%] = 14.9

2. Primary Outcome: Maximum Measured Concentration of BI 1358894 in Plasma
Description: Maximum measured concentration of BI 1358894 in plasma (Cmax). Data presented come from an analysis of variance (ANOVA) model on the logarithmic scale, this model included effects accounting for 'subject' and 'treatment'. The 'subject' effect was considered as random, whereas the 'treatment' effect was considered as fixed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles per Liter
Arm/Group | BI 1358894 | BI 1358894 + Itraconazole
Number analyzed (Participants) | 16 | 16
Nanomoles per Liter | 48.26 (NA) — Geometric standard error = 1.07 | 58.25 (NA) — Geometric standard error = 1.07
Statistical Analysis 1: Comparison: BI 1358894 vs BI 1358894 + Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio = 120.72, 90% CI 2-sided [105.69 to 137.87] — The effect of itraconazole on BI 1358894 is estimated by the ratio of geometric mean (BI 1358894 + itraconazole / BI 1358894). geometric coefficient of variation (gCV) [%] = 21.7

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 to the last quantifiable data point.
  Data presented come from an analysis of variance (ANOVA) model on the logarithmic scale, this model included effects accounting for 'subject' and 'treatment'. The 'subject' effect was considered as random, whereas the 'treatment' effect was considered as fixed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles*Hour per Liter
Arm/Group | BI 1358894 | BI 1358894 + Itraconazole
Number analyzed (Participants) | 16 | 16
Nanomoles*Hour per Liter | 1464.49 (NA) — Geometric standard error = 1.07 | 2686.23 (NA) — Geometric standard error = 1.07
Statistical Analysis 1: Comparison: BI 1358894 vs BI 1358894 + Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio = 120.72, 90% CI 2-sided [105.69 to 137.87] — The effect of itraconazole on BI 1358894 is estimated by the ratio of geometric mean (BI 1358894 + itraconazole / BI 1358894). geometric coefficient of variation (gCV) [%] = 13.3

ADVERSE EVENTS:
Time Frame: For BI 1358894 with the beginning of first administration of BI 1358894 alone + 14 days (336 hours (h)). For itraconazole beginning with the first administration alone up to first administration of BI 1358894 administration in treatment period 2. For the combination with the beginning of administration of BI 1358894 in treatment period 2 + 6 days (144 h) after last administration of itraconazole or 14 days (336 h) after the BI 1358894 administration in treatment period 2, what occurs later.
Description: Treated set (TS): The TS included all subjects who were treated with at least 1 dose of trial drug.
Groups:
- BI 1358894: Oral administration of single dose of 10 milligram (mg) (2 tablets of 5 mg) BI 1358894 with 240 milliliter (mL) of water after an high-fat, high-calorie breakfast on Day 1.
- Itraconazole: Oral administration of 200 mg itraconazole (20 mL of 10 mg/mL solution) with 240 mL of water after an overnight fast for at least 10 hours once daily on Days -3 to 1 until the administration of BI 1358894.
Arm/Group | BI 1358894 | Itraconazole | BI 1358894 + Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 8/16 | 2/16 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1358894 (N=16) | Itraconazole (N=16) | BI 1358894 + Itraconazole (N=16)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 3
Feeling of relaxation (General disorders) | 1 | 0 | 0
Puncture site swelling (General disorders) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 1
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 0 | 4
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT03843151/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT03843151/SAP_001.pdf